CLINICAL TRIAL: NCT02168010
Title: Efficacy and Safety of Analgecine for Low Back Pain: a Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Trial
Brief Title: Analgecine for Treatment of Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VanWorld Pharmaceutical (Rugao) Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: vw1401
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2014-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — neurotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experiment (Experimental): Test Drug Group: 2 times a day; 4 tablets per time (2 tablets of Analgecine and 2 tab. of placebo)
  Interventions: Drug: Analgecine
- PosCtrl (Active Comparator): PosCtrl: Positive Control Group. 2 times a day; 4 tablets / time (2 tab. of Neurotropin and 2 placebo tablets).
  Interventions: Drug: Neurotropin
- Placebo (Placebo Comparator): Placebo Group: 2 times a day; 4 tablets / time (4 placebo tablets).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Analgecine — Analgesic drug under test
  Arms: Experiment
Drug: Neurotropin — Analgesic drug as positive control
  Arms: PosCtrl
Drug: Placebo — Blank tablet as placebo.
  Arms: Placebo

SUMMARY:
The study examines the efficacy and safety of Analgecine in the treatment of chronic pain in patients with low back pain for 3 months after surgical treatment. It is a randomized, placebo-controlled, double blind, multi-center phase III clinical trial. Patients with chronic low back pain for 3 months after surgical treatment is recruited (age between 18 and 70; pain visual analysis scale (VAS) between 3 and 8). After randomization, subjects are divided into 3 groups: 1) Treatment with Analgecine (Experiment group); 2) Treatment with Neurotropin (positive control group); 3) Placebo group. Subjects will be undergone 4 measurement time points on day 0, 7, 14, and 21. In each time points, subjects are required to score their pain with pain VAS and to have regular blood, urine, and renal/liver function tests. The changes of the pain VAS at day 21 are compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain including patients with spinal degeneration, lumbar herniation, lumbar spinal stenosis, and spondylolisthesis
* Pain sustained for 3 or more months after surgical treatment.
* Diagnosis is done by X-ray examination.
* The Visual analysis Scale for Pain is between 3 and 8.

Exclusion Criteria:

* Acute low back pain patients.
* Allergy to the tested drug.
* Patients with tuberculosis, tumors, Cushing's syndrome, endocrine diseases, neuropathic diseases, psychiatric problems, and serious deficit in heart / liver /renal functions.
* Patients with pain caused by vascular diseases, stress, or tumors.
* Patients with pregnancy, lactation, or planning to have pregnancy within 3 months after recruitment.
* Alcoholic and drug addicted subjects
* Dementia patients who can cooperate with the study activities.
* Patients undergone lumber surgery within 3 months at the date of recruitment.
* Patients who are directly related to the research staff.
* Patients who have been participated in other drug clinical trial in the past 3 months at the date of the recruitment.
* Patients who are not fit for the clinical trial based on the research staff observation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change of Visual Analysis Scale on Pain | Day 0, 7, 14 and 21

SECONDARY OUTCOMES:
ECG | Day 0, 21
Routine Hematology Testing | Day 0, 21
Routine Urine Testing | Day 0, 21
Renal / Liver function tests | Day 0, 21
Degree of Improvement of Related Symptoms | Day 0, 7, 14, 21

CONTACTS AND LOCATIONS:
Overall Officials: Steve Chen-Lung Lin, MD, PhD, Study Director — Graduate School of Medicine, Kaohsiung Medical University; Jian Dong, MD, PhD, Principal Investigator — Zhong Shan Hospital, Fudan University
Locations (7):
- China (7):
  - Second Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - No.3 Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shanghai Sixth People's Hosptial, Shanghai, Jiangsu
  - Zhong Shan Hospital, Fudan University, Shanghai, Jiangsu
  - Xijing Hospital, Xi'an, Shaanxi
  - Tiangjin People's Hospital, Tianjin